CLINICAL TRIAL: NCT07280078
Title: Evaluation of a Yoga, Meditation and Mindful Eating Intervention for the Control of Stress, Anxiety, Depression, and Mindfulness in University Students
Brief Title: Yoga, Meditation and Mindful Eating Intervention in University Students
Acronym: Yoga-UDEA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Javier Mauricio Ceballos Rueda, PhD, Universidad de Antioquia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Acta Nº 254 CEI-FE (UDEA)
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-10

CONDITIONS: Stress, Psychological; Anxiety; Depression; Mindfulness; Well-being
Keywords: Yoga, Meditation, Stress, Psychological; Anxiety; Well-being; Mindful Eating; Psychological
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders; Depression | interventions — Yoga; Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga and Meditation Gruop (Active Comparator): University students enrolled in the course "Yoga, Meditation, and Mindful Eating" will participate in a 32-hour holistic intervention. The program integrates theoretical and practical sessions focused on yoga postures (asanas), breathing exercises (pranayamas), meditation, relaxation, and mindful eating practices based on Ayurvedic principles.
  Interventions: Behavioral: Yoga, Meditation, and Mindful Eating

INTERVENTIONS:
Behavioral: Yoga, Meditation, and Mindful Eating — The behavioral intervention combines weekly 2-hour sessions for 16-weeks. Each class includes warm-up exercises, yoga postures for balance and flexibility, breathing techniques (pranayamas), guided meditation, and relaxation. Additionally, participants receive recommendations on healthy habits, conscious nutrition, and physical well-being.

SUMMARY:
The aim of this study is to learn whether a program that combines yoga, meditation, and mindful eating can help reduce stress, anxiety, and depression, and improve mindfulness in university students.

The main questions the study aims to answer are:

* Does participating in yoga, meditation, and mindful eating sessions lower students' levels of stress, anxiety, and depression?
* Does the program improve students' mindfulness and general well-being?

What will happen in the study:

Participants will:

* Attend weekly sessions of yoga, meditation, and mindful eating for 32 hours total.
* Practice physical postures (Asanas), breathing exercises (Pranayama), relaxation, and meditation.
* Receive short lessons about mindful nutrition and healthy lifestyle habits.
* Complete questionnaires before and after the program to measure stress, anxiety, depression, and mindfulness.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students enrolled in the curso "Yoga, Meditation, and Mindful Eating" at the Faculty of Pharmaceutical and Food Sciences (CIFAL), University of Antioquia.
* Willing to participate voluntarily and complete all study assessments.
* Able to attend the full program (32 hours over one academic semester).

Exclusion Criteria:

* Students currently practicing yoga or meditation regularly.
* Pregnant women or participants with any medical condition that prevents safe participation in yoga practice.
* Individuals with severe psychiatric disorders requiring pharmacological treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in academic stress levels measured by the Academic Stress Scale (E-CEA). | Baseline (pre-test, week 1) and after completion of the intervention (post-test, week 16).
  The Academic Stress Scale (E-CEA) evaluates students' perceived academic stress through 54 items assessing methodological, social, and emotional factors related to their studies.

SECONDARY OUTCOMES:
Change in anxiety levels measured by the State-Trait Anxiety Inventory (STAI). | Baseline (pre-test, week 1) and after completion of the intervention (post-test, week 16).
Change in depressive symptoms measured by the Beck Depression Inventory II (BDI-II). | Baseline (pre-test, week 1) and after completion of the intervention (post-test, week 16).

IPD SHARING:
Plan to Share IPD: Yes